CLINICAL TRIAL: NCT01468506
Title: Ultrasound to Predict Steal-Syndrome After Arteriovenous-Fistula Creation (UPSAC - Trial)
Acronym: UPSAC
Status: Withdrawn | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Principal Investigator, Raul Herrera, MD, Director of Clinical Research, Baptist Hospital of Miami, BCVI, Baptist Health South Florida
Other Study IDs: UPSAC version 17 Jul 2011
Record Dates: First submitted 2011-11-03; First posted 2011-11-09 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; arteriovenous fistula
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fistula patients: Consecutive patients with autogenous, brachio-cephalic, brachio-basilic or brachio-brachial arterio-venous fistula creation for hemodialysis

SUMMARY:
The purpose of this study is to analyze and identify pre-, intra-, and post- operative parameters that predict Steal-Syndrome with distal malperfusion after Arterio-Venous Fistulas (AVF) as primary endpoint. Secondary endpoints are pre-, intra-, and post- operative parameters that predict patency and fistula maturation.

DETAILED DESCRIPTION:
This is a prospective study where the research team will acquire data from the patients after they have signed the informed consent form. Data will be collected before, during and after the Arterio-Venous Fistula(AVF)placement, and during follow-up at predefined time intervals:Pre-Operative, Intra-operative, Post-operative, 5-10 days, 4-6 Weeks, 6 Months, and 1 year. These parameters include Digital Brachial Index (DBI) (assessed by Doppler derived brachial artery blood pressure/ photoplethysmographically derived finger blood pressure), flow and pulsatility measurements (derived by duplex ultrasound and pulse volume recording). Assessment of flow and pulsatility will be performed in the artery proximal and distal to the AVF, as well as in the venous outflow. In addition, Demographic parameters and patient comorbidities will be acquired and procedure specific parameters (e.g. location of the fistula) will be documented. During each follow up, clinical evaluation for Steal-Syndrome will be conducted. Steal-Syndrome was defined according to the guidelines of the Society of Vascular Surgery (SVS): Asymptomatic (pulse deficits, doppler signal attenuation, and distal flow reversal) Mild Ischemia: slight coldness and numbness that occurs only during dialysis, may be self-limited, and may resosolve without treatment, and Severe Ischemia: Can be permanent and may be associated with constant pain, severe numbness, digital cyanosis or gangrene, finger contracture, or amputation of a digit hand or forearm. The necessity for and type of re-intervention at the AVF will be documented. Acquisition of data will in no way change the standard of care used in these patients / operations.

Data analysis will be performed after enrolment of 100, 250 and 500 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age
* Autogenous, brachio-cephalic, brachio-basilic or brachio-brachial Arterio- Venous Fistula creation for hemodialysis
* General preoperative requirements for this surgery passed
* Patients willing to adhere to the follow-up
* Patients able to understand and provide informed consent

Exclusion Criteria:

* Less than 18 years of age
* Patient is unable or unwilling to provide consent
* Prosthetic graft creation
* Creation of a radio-cephalic AV-Fistula other than described in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected for this protocol must have the necessity to undergo surgery to receive an Arterio-Venos Fistula (AVF) for hemodialysis in either arm.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Steal-Syndrome | 1 year
  Steal Syndrome as defined according to the guidelines of the Society of Vascular Surgery (SVS): Asymptomatic (pulse deficits, doppler signal attenuation, and distal flow reversal) Mild Ischemia: slight coldness and numbness that occurs only during dialysis, may be self-limited, and may resosolve without treatment, and Severe Ischemia: Can be permanent and may be associated with constant pain, severe numbness, digital cyanosis or gangrene, finger contracture, or amputation of a digit hand or forearm. Standard assessment for steal syndrom at 5-10 days, 4-6 weeks, 6 months, and 1 year.

SECONDARY OUTCOMES:
Time to fistula maturation | 1 year
  Time between fistula creation and time to clinical fistula maturation, standard assessment of fistula maturation at 5-10 days, 4-6 weeks, 6 months, and 1 year
Fistula patency | 1 year
  Time between fistula creation and time to first intervention to restore fistula function (operation, endovascular procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Tsoukas, MD, Principal Investigator — Baptist Hospital Miami, BCVI; Heiko Uthoff, MD, Principal Investigator — Baptist Hospital Miami, BCVI; Philipp Geisbuesch, MD, Principal Investigator — Baptist Hospital Miami, BCVI; Raul Herrera, MD, Study Director — Baptist Hospital of Miami, Baptist Cardiac and Vascular Institute; Barry Katzen, MD, Principal Investigator — Medical Director Baptist Cardiac and Vascular Institute
Locations (1):
- Baptist Hospital of Miami, Baptist Cardiac and Vascular Institute, Miami, Florida, United States